CLINICAL TRIAL: NCT05176925
Title: A Phase II, Open-Label, Single-Arm, Prospective Clinical Study to Investigate the Efficacy and Safety of Tislelizumab Combined With Sitravatinib as Consolidation Treatment in Patients With Locally Advanced, Unresectable NSCLC Who Have Not Progressed Following Definitive, Platinum-based, Concurrent Chemoradiation Therapy
Brief Title: Tislelizumab Combined With Sitravatinib as Consolidation Treatment Following Concurrent Chemoradiation in Patients With Locally Advanced, Unresectable NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated per sponsor recommendation
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2111245-17
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; sitravatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with sitravatinib (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Sitravatinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg IV D1, Q3W
Drug: Sitravatinib — The starting dose of sitravatinib in this study is 70 mg, oral once daily. After receiving 2 cycles of starting dose at 70 mg once daily with sitravatinib, if patients were tolerated well with study treatment (without AEs definitely related to sitravatinib nor TRAEs leading to sitravatinib dose reduction and interruption), it is recommended to escalate sitravatinib dose to 100 mg once daily at the discretion of the investigators after discussion with patients.

SUMMARY:
This study aims to evaluate the 1-year progression free survival (PFS) rate of tislelizumab combined with sitravatinib as assessed by investigators per RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status≤1.
* Life expectancy ≥ 3 months.
* Eligible patients for this study must have locally advanced, Stage III NSCLC that is considered unresectable. histologically- or cytologically-documented NSCLC who present with locally advanced, unresectable (Stage III) disease (according to Version 8 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology). Patients must not have progressed following definitive, platinum-based, concurrent chemoradiation therapy.
* First dose of study treatment is no later than 42 days after cCRT.
* Adequate organ function as indicated by the following laboratory values (obtained ≤ 7 days before first dose)

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L,
  2. Platelets ≥ 100 × 10^9/L,
  3. Hemoglobin ≥ 90 g/L.
  4. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x upper limit of normal (ULN).
  5. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
  6. Serum total bilirubin ≤ 1.5 x ULN.
  7. Aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 x ULN.
  8. Serum albumin ≥25 g/L（2.5 g/dL).
  9. Serum creatinine ≤ 1.5 x ULN or estimated glomerular. filtration rate (GFR) >50 mL/min by Cockcroft-Gault equation.
* Able to provide written informed consent by the patient or by the patient's legally acceptable representative and can understand and agree to comply with the requirements of the study.
* Patients of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drugs.

Exclusion Criteria:

* Mixed small cell and non-small cell lung cancer histology.
* Received prior anti-VEGF mAb or VEGFR TKI agents and prior therapies targeting PD-1, PD-L1, CTLA-4 or other immune checkpoints.
* Have any unresolved AE≥Grade 2 from prior cCRT，radiotherapy induced hearing loss, hair loss, peripheral sensory neuropathy and fatigue is excluded.
* Grade ≥2 radiation pneumonitis while receiving cCRT.
* Patients with known EGFR mutation, or ALK or ROS1 rearrangement.
* Treatment with any approved systemic anti-cancer therapy or systemic immune-stimulatory agents (including but not limited to interferons, interleukin IL-2, and tumor necrosis factor) within 4 weeks prior to initiation of study treatment.
* Administration of live vaccine ≤ 4 weeks before the first dose of study treatment.
* History of allergic reactions to any study drugs.
* Patients with untreated chronic hepatitis B (HBV) or chronic HBV carriers whose HBV DNA ≥ 500 IU/mL, patients with active hepatitis C (HCV).
* Active autoimmune diseases that require treatment and may affect study treatment estimated by investigator.
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or any other immunosuppressive medication≤ 14 days before first dose of study drugs that may affect study treatment estimated by investigator.
* Severe chronic or active infections requiring systemic antibacterial, antifungal, within 14 days prior to first dose of study drug(s).
* Prior allogeneic stem cell transplantation or organ transplantation.
* Any of the following cardiovascular risk criteria:

  1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of study drugs.
  2. Symptomatic pulmonary embolism ≤ 28 days before first dose of study drugs.
  3. Any history of acute myocardial infarction ≤ 6 months before first dose of study drugs.
  4. Any history of heart failure meeting New York Heart Association Classification III or IV ≤ 6 months before first dose of study drugs.
  5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of study drugs.
  6. Any history of cerebrovascular accident ≤ 6 months before first dose of study drugs.
  7. QTc interval (corrected by Fridericia's method) > 450 msec (for males)/ > 470 msec (for females). Note: If QTc interval is > ULN on initial ECG, a follow up ECG will be performed to exclude result.
  8. Current left ventricular ejection fraction (LVEF) < institutional LLN as assessed by echocardiography (ECHO).
  9. Any episode of syncope or seizure ≤ 28 days before the first dose of study drug(s).
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg).
* Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring within 6 months before first dose of study drugs.
* Regardless of the severity, patients with any signs or medical history of bleeding; within 4 weeks prior to allocation, patients with any bleeding events ≥ CTCAE level 3, unhealed wounds, ulcers, or fractures.
* Hemoptysis>50ml/d.
* With central cavitation or tumor shown by imaging to be located around important vascular structures or if the investigator determines that the tumor is likely to invade important blood vessels and may cause fatal bleeding.
* Inability to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Patients requiring treatment with gastric pH-modifying medications including proton pump inhibitors and/or H2 antagonist medications. Patients may switch to use of antacids.
* History of uncontrolled diabetes, hypertension, pulmonary fibrosis, acute lung diseases, etc.
* Significant history or clinical manifestation of any organ systems disorder, as determined by the investigator.
* Any major surgical procedure requiring general anesthesia≤28 days before initiation of study treatment.
* Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that would be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
* Known history of HIV infection.
* Any active malignancy≤2 years before first dose of study treatment except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
* Pregnant or breastfeeding woman.
* Concurrent participation in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
1-year Progression-Free-Survival (PFS) rate assessed by investigators per RECIST 1.1 | Start of treatment until 1-year follow-up
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.

SECONDARY OUTCOMES:
PFS (Progression-Free-Survival) | Up to 4 years
  From date of treatment start until the date of progression or the date of death due to any cause, evaluated according to RECIST 1.1 criteria,
Objective Response Rate (ORR) | Up to 4 years
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DOR) | Up to 4 years
  Duration of response is defined as the time from first documented response of CR or PR to date of first documented progression or death, according to RECIST 1.1 criteria
DCR (Disease Control Rate) | Up to 4 years
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD), evaluated according to RECIST 1.1 criteria.
OS (Overall Survival) | From date of treatment start until the date of death from any cause or censored at the last day that the subjects are documented to be alive, whichever came first, assessed up to 4 years.
  From date of treatment start to any cause death or last follow-up.
Time to Distant Metastasis (TTDM) | Up to 4 years.
  From date of treatment start to distant metastasis.
Adverse events (per CTCAE v5.0 criteria) | Up to 4 years
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of adverse events (AEs) and serious adverse events (SAEs) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China